CLINICAL TRIAL: NCT00760123
Title: Lymphedema Prevention in Breast Cancer: a Simple Blind, Randomized, Prospective Clinical Trial of the Efficacy of Physical Therapy
Brief Title: Lymphedema Prevention in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Maria Torres Lacomba, PhD, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ID1124
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: BREAST CANCER; LYMPHEDEMA
Keywords: Lymphedema; Prevention; Breast cancer; Physical therapy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early Physical Therapy including a manual lymph-drainage technique, progressive massage of the scar, and progressive active and action-assisted shoulder exercises started in conjunction with functional activities and proprioceptive neuromuscular facilitation without resistance and educational strategy including instruction with printed materials about the lymphatic system, concepts of normal load versus overload, lymphedema source, the identification of possible precipitating factors, etc.
  Interventions: Other: Early Physical Therapy and Educational strategy
- 2 (Other): Educational Strategy: instruction with printed materials about the lymphatic system, concepts of normal load versus overload, lymphedema source, the identification of possible precipitating factors, etc.
  Interventions: Other: Early Physical Therapy and Educational strategy

INTERVENTIONS:
Other: Early Physical Therapy and Educational strategy — Experimental group:
  physical therapy including a manual lymph-drainage technique, progressive massage of the scar, and progressive active and action-assisted shoulder exercises started in conjunction with functional activities and proprioceptive neuromuscular facilitation without resistance and Educational strategy including instruction with printed materials about the lymphatic system, concepts of normal load versus overload, lymphedema source, the identification of possible precipitating factors,etc.
  Other: control group: only the educational strategy

SUMMARY:
OBJECTIVE: To find out the effectiveness of early application of physical therapy in the prevention of lymphedema after breast surgery and lymphadenectomy.

DESIGN: Randomized, controlled and single blinded clinical trial. Three years duration. Patients will be randomly assigned to one of these groups: Experimental group: Early physical therapy + training in means of prevention; Control group: just training in means of prevention. In both groups several physical therapy assessments will be undertaken: 1st before surgery; 2nd immediately after surgery; 3rd after completing intervention; 4th, 5th and 6th after 3, 6, 12 and 24 months.

SUBJECTS: Women with breast cancer treated with breast surgery including lymphadenectomy in Principe de Asturias Hospital, provided that there is no contraindication for physical therapy, and after reading, understanding and freely signing an informed consent form.

SAMPLE SIZE: A total of 116 subjects will be included in the study (58 subjects in each group), assuming a 15% of drop-outs and at least 20% reduction, with a statistical power of 60%.

DATA ANALYSIS: To find out the effectiveness of intervention we will compare the rate of lymphedema in both groups by means of a logistic regression analysis, in which the main factor is the intervention group. Other factors aimed to control the effect of the intervention will also be included. In order to compare the rate of appearance of lymphedema in both groups, a survival analysis will also be included.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive women diagnosed with breast cancer and undergoing unilateral surgery with axillary lymph-node dissection at the Príncipe de Asturias Hospital in Alcalá de Henares, Madrid (Spain) are candidates for inclusion in the study.

Exclusion Criteria:

* Patients without axillary lymph-node dissection or with bilateral BC, systemic disease, locoregional recurrence, or any contraindication to physical therapy are excluded from the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-05; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Circumference measurements of the upper limbs using at 5 cm intervals from the elbow fold preoperatively prior to randomization and then post-operatively on hospital discharge (between Day 3 and Day 5), 4 weeks, and 3, 6, 12 and 24 months after surgery. | 2 years

SECONDARY OUTCOMES:
Pain, measured using the Visual Analogue Scale and Shoulder abduction measured using a digital goniometer. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: María Torres Lacomba, Prof., Principal Investigator — Alcalá University; Maria José Yuste Sánchez, Prof., Study Chair — Alcalá University; Álvaro Zapico Goñi, MD, Study Chair — Principe de Asturias Hospital University; David Prieto Merino, Study Chair — Department of Epidemiology and Population Health, London School of Hygiene & Tropical Medicine, UK; Orlando Mayoral del Moral, Prof., Study Chair — Provincial Hospital.
Locations (2):
- Spain (2):
  - Alcalá University, Alcalá de Henares, Madrid
  - María Torres Lacomba, Alcalá de Henares, Madrid

REFERENCES:
- [Background] Stout Gergich NL, Pfalzer LA, McGarvey C, Springer B, Gerber LH, Soballe P. Preoperative assessment enables the early diagnosis and successful treatment of lymphedema. Cancer. 2008 Jun 15;112(12):2809-19. doi: 10.1002/cncr.23494. PMID 18428212